CLINICAL TRIAL: NCT00874068
Title: The Effects of Dietary Palmitic Acid Triacylglyceride Position on Anthropometric Measures, Bone Strength Parameters, Stool Characteristics and Stool Biochemistry in Preterm and Term Infants
Brief Title: The Effects of Dietary Palmitic Acid Triacylglyceride Position on Bone Strength Parameters in Infants
Acronym: InFat_002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Fabiana Bar-Yoseph, Enzymotec
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PAL1
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Personal Satisfaction
Keywords: term infants; preterm infants; bone strength; Speed of sound (SOS); Ultrasound
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard vegetable oil formula (Active Comparator)
  Interventions: Other: Standard vegetable oil based infant formula
- InFat (Active Comparator)
  Interventions: Other: InFat™ based infant formula
- Breast-fed (No Intervention)

INTERVENTIONS:
Other: InFat™ based infant formula — high sn-2 palmitic acid oil based infant formula
  Other Names: high sn-2 palmitic acid; structured triglyceride
  Arms: InFat
Other: Standard vegetable oil based infant formula — standard vegetable oil based infant formula
  Other Names: standard vegetable oil
  Arms: Standard vegetable oil formula

SUMMARY:
The purpose of this study is to determine the effect of high sn-2 palmitic acid based infant formula on bone strength parameters.

DETAILED DESCRIPTION:
InFatTM is an advanced basic-fat ingredient, which mimics the fat composition and properties of human milk fat and enabling optimal intake of the essential calcium and energy (in the form of fatty acids) and easy digestion. These benefits are the results of a unique fatty acid composition on the glycerol backbone, which ensure high level of palmitic acid at the middle (sn-2) position.

The purpose of this study is to determine the effect of high sn-2 palmitic acid based infant formula on bone strength parameters, anthropometric parameters, wellbeing and stool characteristics in term and preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age above 32 weeks as determined by menstrual history and corroborated by prenatal US and/or physical examination.
2. Birth weight appropriate for gestational age (AGA) using current CDC growth charts, and above 1750gr.
3. The mother had unequivocally decided not to breast-feed (in formula groups) or the mother had decided to breast feed (in human breast milk group).
4. The infant is apparently healthy.
5. Parental/ legal guardian written inform consent
6. Apgar after 5 minutes >7
7. Enrolled within their first 14 days of life for term infants and first month of life for preterm infants
8. At enrollment: clinical stability and acceptable weight gain

Exclusion Criteria:

1. The infant suffer from a congenital or chromosomal disorder (Cystic fibrosis, Tracheomalacia, Tracheoesophageal fistula, major congenital heart disease, down-syndrome)
2. The infant suffer from neonatal morbidities:

   * Bronchopulmonary dysplasia (BPD)
   * Intraventricular Hemorrhage3-4 (IVH)
   * Necrotizing Enterocolitis (NEC)
3. Laboratory or clinical sings of Osteopenia
4. The infant suffers from any suspected or known metabolic or physical limitations interfering with feeding or normal metabolism (require a special formula)
5. The mother suffers from any disease or disability that may interfere with her ability to take care of her infant
6. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
bone strength parameters | baseline, 40 corrected gestation weeks, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
stool characteristics | baseline, 40 corrected gestation weeks, 6 weeks, 12 weeks
Antropometric measurements | baseline, 40 corrected gestation weeks, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Derived] Litmanovitz I, Bar-Yoseph F, Lifshitz Y, Davidson K, Eliakim A, Regev RH, Nemet D. Reduced crying in term infants fed high beta-palmitate formula: a double-blind randomized clinical trial. BMC Pediatr. 2014 Jun 19;14:152. doi: 10.1186/1471-2431-14-152. PMID 24942975